CLINICAL TRIAL: NCT00108654
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Booster Dose of a Recombinant Multiclade HIV-1 Adenoviral Vector Vaccine, VRC-HIVADV014-00-VP, in Uninfected Subjects Who Where Previously Immunized With VRC-HIVDNA016-00-VP in VRC 00
Brief Title: Vaccine Treatment for HIV-Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050140; 05-I-0140
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-01-15

CONDITIONS: Healthy
Keywords: HIV-Negative; Healthy; Immunity; Preventive; Virus; Healthy Volunteer
MeSH Terms: conditions — Virus Diseases

INTERVENTIONS:
Drug: VRC-HIVADV014-00-VP

SUMMARY:
This study will determine the safety and side effects of an experimental adenoviral vector vaccine given to patients who previously received a different HIV vaccine (VRC-HIVDNA016-00-VP) in a prior NIAID study. The study will also monitor participants for the social impact of being in an HIV vaccine study (e.g., problems with insurance, health care, friends, family, employment, housing, and so forth). The study vaccine is made using an adenovirus (a common virus that causes upper respiratory infections, such as the common cold, eye infection, urine infection or diarrhea) that has been modified to contain DNA that codes for three HIV proteins. The modified virus cannot reproduce in the body and cannot cause HIV disease or adenoviral infections.

Healthy volunteers who previously received three injections of the VRC-HIVDNA016-00-VP under the NIAID study VRC 007 (protocol 04-I-0254) may be eligible for this study.

Participants receive one injection of the adenoviral vector vaccine. It is given the day they enroll in the study, as a single injection in an upper arm muscle. Also on that day they have a brief physical examination, medical history, blood and urine tests, pregnancy test for women, and counseling, as needed, about HIV and pregnancy avoidance. Subjects are observed for side effects for at least 30 minutes after the vaccination and are required to telephone the clinic staff 1 to 2 days after the injection for follow-up. In addition, they are given a diary card to take home, on which they record their temperature and any symptoms daily for 5 days.

Subjects return to the clinic for 5 follow-up visits at weeks 2, 4, 6, 12 and 24 after the injection. At each visit they are checked for health changes or problems since the last visit, asked how they are feeling and what medications they are taking. They have blood drawn at every visit and urine samples collected at most visits. They are tested for HIV three or more times and are questioned about their sexual behavior and drug use. They also complete a "social impact" questionnaire at the last visit.

Subjects are asked to undergo apheresis at the week 4 visit. This procedure allows collection of a larger number of white blood cells than can be obtained by a simple blood draw. The white cells are studied to see how the immune system responds to the study vaccine. For apheresis, blood is collected through a needle in an arm vein and spun in a machine that separates the components. The white blood cells are extracted and the rest of the blood is returned to the body through the same needle. Subjects who do not undergo apheresis have about 1/3 cup of blood sample drawn using a needle.

DETAILED DESCRIPTION:
Study Design: This is a Phase I open-label study to examine safety, tolerability and immune response of a multiclade HIV adenoviral vector vaccine as a booster vaccination in uninfected adults. The hypothesis is that this vaccine will be safe as a booster vaccine and elicit immune responses to HIV. The primary objective is to evaluate the safety and tolerability of a VRC-HIVADV014-00-VP booster vaccination in uninfected subjects who previously received 3 injections of VRC-HIVDNA016-00-VP. The secondary objectives include immunogenicity evaluations, adenovirus serotype 5 (Ad5) antibody titers, and social impacts. Exploratory evaluations include epitope mapping and other immunogenicity evaluations.

Product Description: VRC-HIVADV014-00-VP (rAd) is a recombinant product composed of 4 adenoviral vectors (in a 3:1:1:1 ratio) that encode the HIV-1 Gag/Pol polyprotein from clade B and HIV-1 Env glycoproteins from clades A, B, and C, respectively.

Subjects: Healthy adult volunteers who previously received three injections of VRC-HIVDNA016-00-VP at a dosage of 4 mg in the VRC 007 study (04-I-0254). The subjects in these groups were between 20 and 36 years old at time of enrollment in VRC 007; those who participate in VRC 010 will be no more than 36 weeks older at the time of enrollment into VRC 010.

Study Plan: Up to fourteen volunteers will receive one 1 mL injection of the study agent at a dosage of 1010 particle units (PU) intramuscularly (IM) in a deltoid muscle. Safety and immunogenicity will be evaluated by follow-up visits over the subsequent 24 weeks. The peripheral blood mononuclear cell (PBMC) sample for immunogenicity studies collected at Week 4 after vaccination will be obtained by apheresis if the subject is willing and eligible for apheresis and an apheresis appointment can be conveniently scheduled in the interval specified; otherwise PBMCs will be obtained from 80 mL blood collected by phlebotomy.

Study Duration: Subjects will be evaluated at 6 or more clinical visits for 24 weeks after the study injection.

Study Endpoints: The primary endpoint is safety of the vaccine administered at a dose of 10(10) PU by IM injection. Secondary endpoints are immunogenicity as indicated by HIV-specific antibody through Week 4, cellular immune responses through Week 6, Ad5 antibody titer at Week 0 and Week 4 and social impact at Week 24. Exploratory analyses include immunogenicity at Weeks 12 and 24, Ad5 antibody titer at Week 24 and epitope mapping of the CD8+ and CD4+ T cell responses at Week 4.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

Enrolled into VRC 007 no more than 36 weeks prior to VRC 010 enrollment and completed three injections of 4 mg of study vaccine in VRC 007 (04-I-0254) without experiencing a serious adverse event (SAE) that was possibly, probably or definitely related to study vaccine.

Available for clinical follow-up for 24 weeks after enrollment into VRC 010.

Completion of an Assessment of Understanding prior to enrollment and able to verbalize understanding of all questions answered incorrectly.

Able and willing to complete the informed consent process.

Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.

Willing to donate blood for sample storage to be used for future research.

Willing to discuss HIV infection risks and amenable to risk reduction counseling.

In good general health without clinically significant medical history and satisfactory completion of the screening process.

Laboratory Criteria within 28 days prior to enrollment:

Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to13.5 g/dL for men;

WBC = 3,300-12,000 cells/mm(3);

Differential either within institutional normal range or accompanied by site physician approval;

Total lymphocyte count greater than or equal to 800 cells/mm(3);

Platelets = 125,000 - 550,000/mm(3);

ALT (SGPT) less than or equal to 1.25 x upper limit of normal;

Serum creatinine less than or equal to 1 x upper limit of normal (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males);

Normal urinalysis defined as negative glucose, negative or trace protein, and no clinically significant blood in the urine;

Negative HIV PCR (i.e., less than the lower limit of detection or less than 50 RNA copies/mL);

Negative Hepatitis B surface antigen;

Negative anti-HCV (hepatitis C virus antibody) and negative HCV PCR.

Female-Specific Criteria:

Negative beta-HCG pregnancy test (urine) on day of study enrollment for women presumed to be of reproductive potential.

A female participant must meet one of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 24 of the study,

or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 24 of the study by one of the following methods:

condoms, male or female, with or without a spermicide;

diaphragm or cervical cap with spermicide;

intrauterine device;

contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method;

male partner has previously undergone a vasectomy for which there is documentation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

Women:

Breast-feeding or planning to become pregnant during the 24 weeks of study participation.

Volunteer has received any of the following substances:

Immunosuppressive or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis).

Blood products within 120 days prior to HIV screening.

Immunoglobulin within 60 days prior to HIV screening.

Live attenuated vaccines within 30 days prior to initial study vaccine administration.

Investigational research agents within 30 days prior to study vaccine administration.

Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration.

Current anti-TB prophylaxis or therapy.

Volunteer has a history of any of the following clinically significant conditions:

Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain.

Autoimmune disease or immunodeficiency.

Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.

Diabetes mellitus (type I or II), with the exception of gestational diabetes.

History of thyroidectomy or thyroid disease that required medication within the past 12 months.

Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.

Hypertension that is not well-controlled by medication or is more than 145/95 at enrollment.

Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.

Syphilis infection that is active or a positive serology due to a syphilis infection treated less than six months ago.

Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.

Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.

Asplenia or any condition resulting in the absence or removal of the spleen.

Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to enrollment, history of a suicide plan or attempt.

Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 20 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14
Dates: Start 2005-04-13; Study Completion 2008-01-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Pantaleo G, Demarest JF, Soudeyns H, Graziosi C, Denis F, Adelsberger JW, Borrow P, Saag MS, Shaw GM, Sekaly RP, et al. Major expansion of CD8+ T cells with a predominant V beta usage during the primary immune response to HIV. Nature. 1994 Aug 11;370(6489):463-7. doi: 10.1038/370463a0. PMID 8047166
- [Derived] Koup RA, Roederer M, Lamoreaux L, Fischer J, Novik L, Nason MC, Larkin BD, Enama ME, Ledgerwood JE, Bailer RT, Mascola JR, Nabel GJ, Graham BS; VRC 009 Study Team; VRC 010 Study Team. Priming immunization with DNA augments immunogenicity of recombinant adenoviral vectors for both HIV-1 specific antibody and T-cell responses. PLoS One. 2010 Feb 2;5(2):e9015. doi: 10.1371/journal.pone.0009015. PMID 20126394